CLINICAL TRIAL: NCT06137768
Title: A Trial to Evaluate the Efficacy and Safety of HRS-5965 Tablets in Primary IgA Nephropathy
Brief Title: A Trial of HRS-5965 Tablets in Primary IgA Nephropathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5965-201
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group A: HRS-5965; high dose (Experimental)
  Interventions: Drug: HRS-5965
- Treatment group B: HRS-5965; medium dose (Experimental)
  Interventions: Drug: HRS-5965
- Treatment group C: HRS-5965; low dose (Experimental)
  Interventions: Drug: HRS-5965
- Treatment group D: Placebo. (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment group E (Experimental)
  Interventions: Drug: HRS-5965

INTERVENTIONS:
Drug: HRS-5965 — HRS-5965
  Arms: Treatment group A: HRS-5965; high dose; Treatment group B: HRS-5965; medium dose; Treatment group C: HRS-5965; low dose; Treatment group E
Drug: Placebo — Placebo.
  Arms: Treatment group D: Placebo.

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HRS-5965 tablets for primary IgA nephropathy. To explore the effective dosage of HRS-5965 tablets for primary IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent；
2. Weight ≥35 kg, Body mass index (BMI) < 37.5kg /m2;
3. Primary IgA nephropathy was confirmed by renal biopsy within 5 years;
4. 24-UPE≥ 0.75g /24h, or UPCR≥ 0.8g/g at screening and prior to randomization;
5. eGFR≥30 ml/min/1.73m2 at screening and prior to randomization; (CKD-EPI formula)
6. A fertile female subject or a male subject whose partner is a fertile female, who has not had a fertility, sperm/egg donation plan from the signing of the informed consent to 1 month after the last dose, and voluntarily takes effective contraceptive measures (including the partner);
7. Receiving optimal supportive therapy including RAS blockers for 12 weeks and stabilizing the dose for at least 4 weeks after reaching the maximum recommended dose or the maximum tolerated dose prior to randomization;

Exclusion Criteria:

1. Allergic to any RAS blockers, investigational products, or components as evaluated by the investigator;
2. Patients with secondary IgA nephropathy as determined by the investigator;
3. IgA nephropathy with rapid decline of renal function; Kidney pathology indicated that more than 50% of the glomerulus had large crescent body formation, which may affect the study results; Tubule atrophy - interstitial fibrosis of more than 50%;
4. Patients with a history of immunodeficiency disease; Or in combination with other systemic diseases likely to cause proteinuria;
5. Have any organ transplant;
6. Patients with chronic recurrent infections within 1 year prior to screening, such as liver abscess and pyelonephritis; Or subjects with active infection who requiring intravenous antibiotic therapy within 2 weeks prior to randomization;
7. Patients with a history of malignant neoplasms;
8. Patients with a history of severe trauma or major surgery within 12 weeks prior to screening, or who plan to undergo surgery during the study period;
9. Patients with a history of blood donation or a history of severe blood loss (≥400 mL blood loss) within 12 weeks prior to screening, or who have received blood transfusions within 12 weeks prior to screening;
10. The presence of a disease or medical condition determined by the investigator might affect drug absorption, distribution, metabolism, and excretion;
11. As determined by the investigator, the subject has any of the following: progression or recovery of a disease;
12. Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), or total bilirubin exceeding 3 times the upper limit of normal (ULN) at screening;
13. Participants who have participated in a clinical trial of any drug or medical device within 12 weeks prior to randomization and are expected to have residual effects of the investigational treatment (as determined by the investigator), or who were within the follow-up period of a clinical study, or within 5 half-lives of the investigational drug, or within 30 days (whichever is older) before screening;
14. Women who are pregnant or breastfeeding;
15. A history of drug abuse;
16. Any physical or mental illness or condition that, as determined by the investigator, is likely to increase the risk of the study, affect the subject's adherence to the protocol, or prevent the subject from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Ratio of 24-hour Urinary protein to creatinine ratio (UPCR) to baseline | Baseline and Week 12

SECONDARY OUTCOMES:
Ratio of 24-hour Urinary protein to creatinine ratio (UPCR) to baseline | Baseline and Week 24
Ratio of 24-hour Urinary protein to creatinine ratio (UPCR) to baseline | up to Week 24
Ratio of 24-hour Urinary protein excretion（UPE） to baseline | up to Week 24
Change from baseline of estimated glomerular filtration rate（eGFR） | up to Week 24
Change from baseline of serum creatinine | up to Week 24
Ratio of Urinary protein to creatinine ratio and Urinary albumin to creatinine ratio to baseline | up to Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639